CLINICAL TRIAL: NCT00740194
Title: Reciprocal Influence of Sex Steroid Environment and Adipocyte Function in Men.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007/279
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: Physiology; males
MeSH Terms: interventions — Aromatase Inhibitors; Estradiol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Aromatase inhibition
  Interventions: Drug: Aromatase inhibition
- 2 (Active Comparator): Estradiol
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Aromatase inhibition — Letrozole
  Arms: 1
Drug: Estradiol — Dermestril
  Arms: 2

SUMMARY:
Aromatase inhibition versus estradiol during 1 week

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained.
* Male subjects
* Age 18 - 40
* weight < 120 kg

Exclusion Criteria:

* Primary hypogonadism or secondary hypogonadism due to genetic causes (Kallman syndrome etc.), tumors, infiltrative diseases, infections, pituitary apoplexy, trauma, critical illness, chronic systemic illness or intentional.
* Treatment with insulin, corticoids, opiates (on a daily basis), androgen- or estrogen analogs or CYP2A6 substrates (Dexmedetomidine, Ifosfamide, Methoxsalen, Miconazole, Tranylcypromine).
* Impaired renal function defined as serum-creatine > 1.5 mg/dL
* Impaired liver function, defined as ALAT > 2.5 times upper limit of normal
* Clinically significant active cardiovascular disease including history of myocardial infarction within the past 6 months and/or heart failure (NYHA class III or IV) at the discretion of the investigator
* Cancer or any clinically significant disease or disorder, which in the investigator's opinion could interfere with the results of the trial
* Palpable prostate nodule or induration, PSA > 3 ng/mL, prostatism, untreated sleep apnee syndrome, erythrocytosis (hematocrit > 50%) or hyperviscosity.
* Known or suspected abuse of alcohol or narcotics
* Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Effects of sex steroids on adipocytes | 1 week

SECONDARY OUTCOMES:
Effects of sex steroids on lipid metabolism | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Ruige, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be